CLINICAL TRIAL: NCT04839055
Title: The Purpose of This Study is to Compare the Therapy Effects and Clinical Safety of a Regulatory Metabolic Compound, Coenzyme A (CoA) With a Marketed Drug, Abiraterone, in Chinese Patients With Castration-resistant Prostate Cancer (CRPC) .
Brief Title: The Effects of Coenzyme A Combined With Abiraterone on Patients With CRPC
Acronym: CoA-CRPC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangnan University (Other)
Collaborators: Affiliated Hospital of Jiangnan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JiangnanU RWang-1
Record Dates: First submitted 2021-04-08; First posted 2021-04-09 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Castration-resistant Prostate Cancer
MeSH Terms: interventions — abiraterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Coenzyme A 200U (Experimental): Coenzyme A 200U per day
  Interventions: Drug: Coenzyme A Combined With Abiraterone
- Placebo Comparator: Placebo (Placebo Comparator): Abiraterone without coenzyme A
  Interventions: Drug: Abiraterone

INTERVENTIONS:
Drug: Coenzyme A Combined With Abiraterone — Abiraterone 4 pieces per day. Coenzyme A 200U
  Arms: Experimental: Coenzyme A 200U
Drug: Abiraterone — Abiraterone
  Arms: Placebo Comparator: Placebo

SUMMARY:
The purpose of this study is to compare the therapy effects and clinical safety of a regulatory metabolic compound, coenzyme A (CoA) with a marketed drug, abiraterone, in Chinese patients with castration-resistant prostate cancer (CRPC) .

DETAILED DESCRIPTION:
Prostate Cancer (PCa) has developed into the second most common cancer in men. In The United States, PCa has the highest morbidity in man. In China, the incidence rate is lower than in Europe and the US, but it is growing faster and faster. Androgen deprivation therapy (ADT) has been the most commonly used treatment for men with advanced prostate cancer for hundreds of years, effective in more than 85 percent of cases, but usually after 20 months or so, half of patients will inevitably develop castration-resistant prostate cancer (CRPC), which will become resistant to ADT, and patients will relapse. There are several treatments that are trying to address this problem. Such as the chemotherapy docetaxel, cabataxel, and the radioactive drug radium 223 dichloride; PARP inhibitor olaparib, but the efficacy is limited.

For finding some new pathways and targets to treat CRPC, a model of PCa persister cell was first been established at a cellular level in this study. In light of the new target, we first find a being used clinically drug, Coenzyme A (CoA), through prescription sieve to treat enzalutamide or abiraterone drug-fast CRPC patients. CoA functions as an acyl group carrier and assists in transferring fatty acids from the cytoplasm to mitochondria. It is also involved in the oxidation and catabolism of fatty acids. There is an efficient drug action at a cellular level and in animals, and we look forward to it at clinical utility.

ELIGIBILITY:
Inclusion Criteria:

- 18-100 years of age combined use with abiraterone or enzalutamide CRPC

Exclusion Criteria:

- pregnancy acute liver disease or hepatic dysfunction, as determined by levels of alanine aminotransferase (ALT) or aspartate aminotransferase levels (AST) more than 2-fold the upper normal limit nephrotic syndrome or serum creatinine (Cr) ≥2-fold the upper normal limit and creatine phosphokinase (CK) more than 3-fold the upper normal limit primary hypothyroidism psychiatric patients poorly controlled hypertension, as indicated by a Systolic Blood Pressure >180 mmHg or Diastolic Blood Pressure >110 mmHg using contraceptive agent using immunosuppressive drugs, prohibited medication or other non-PCa drugs long-term using CoA drug

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-03-18 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Total prostate specific antigen (TPSA) level | 2 weeks
  The primary efficacy variable from 12.82 ng/mL to 13.01 ng/mL in serum TPSA level and 2 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: YongQuan Chen, MD, Study Chair — Jiangnan University
Locations (1):
- Jiangnan University, Wuxi, Jiangsu, China